CLINICAL TRIAL: NCT00503802
Title: Turbinate Reduction & CPAP Use: A Randomized Blinded OSA (TURBO) Trial
Brief Title: Randomized Clinical Trial of Nasal Turbinate Reduction to Improve Continuous Positive Airway Pressure (CPAP) Outcomes for Sleep Apnea
Acronym: TURBO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Ed Weaver, Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 30678-D; 06-3050-D 02 (Other: University of Washington Human Subjects Division); R01HL084139 (NIH)
Record Dates: First submitted 2007-07-17; First posted 2007-07-19 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2013-06

CONDITIONS: Sleep Apnea Syndromes; Nasal Obstruction; Turbinate Hypertrophy
Keywords: Sleep Apnea; Sleep disordered breathing; Nasal Obstruction; Turbinate; Radiofrequency; Continuous positive airway pressure; CPAP; Sleep surgery
MeSH Terms: conditions — Sleep Apnea Syndromes; Nasal Obstruction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Active RF treatment
  Interventions: Procedure: Radiofrequency Turbinate Reduction
- 2 (Sham Comparator): Sham RF treatment
  Interventions: Procedure: Sham RF

INTERVENTIONS:
Procedure: Radiofrequency Turbinate Reduction — Radiofrequency Turbinate Reduction
  Arms: 1
Procedure: Sham RF — The steps of the procedure are as follows: 1) application of topical anesthetic to the turbinate mucosa bilaterally; 2) injection of 1.0 ml of lidocaine 1% with epinephrine 1:100,000 with a 30-gauge needle into each inferior turbinate anteriorly; 3) delay five minutes for local anesthetic to take full effect; 4) re-insertion of the anesthetic needle to check for complete anesthesia on one side, and injection of another 1.0 ml of lidocaine 1% with epinephrine 1:100,000 5) placement of the radiofrequency electrode (23-gauge, 1 cm long) into the inferior turbinate; 6) delivery of 300 Joules of radiofrequency energy to the turbinate over 29 seconds (no energy will be delivered in sham procedure)7) placement of a cotton pledget (soaked in oxymetazoline solution 0.05%) against the treatment site 8) repeat steps 3 - 8 for the contra-lateral inferior turbinate; 9) removal of the cotton pledgets after several minutes; and 11) observation of hemostasis.
  Arms: 2

SUMMARY:
Obstructive sleep apnea occurs in 2-4% of middle age adults and results in significant morbidity and mortality. The first line therapy is provision of continuous positive airway pressure (CPAP) via a nasal mask chronically. Nasal resistance related to nasal turbinate enlargement may compromise CPAP treatment. This randomized double-blind sham-placebo-controlled trial tests the hypothesis that nasal turbinate reduction improves the nasal passage, CPAP use, and sleep apnea quality of life in newly diagnosed sleep apnea patients who are recommended CPAP therapy.

DETAILED DESCRIPTION:
Obstructive sleep apnea syndrome afflicts at least 2 - 4% of adults and is associated with significant morbidity and mortality. Continuous positive airway pressure (CPAP) therapy is the primary treatment for sleep apnea in adults, but non-adherence to CPAP limits its effectiveness. Even with maximal medical therapy, nasal obstruction is common in sleep apnea patients and may hamper both CPAP adherence and efficacy. However, the most common cause of nasal obstruction in sleep apnea patients (turbinate hypertrophy) is surgically correctable. Treatment of nasal obstruction may lead to more successful use of CPAP. The long-term goal of the proposed research is to develop a novel, multi-disciplinary, multi-modal approach to therapy, in order to improve clinically important treatment outcomes for sleep apnea. The short-term objectives of this proposal are to:

1. Quantify the effect of nasal turbinate reduction on the nasal airway;
2. Determine whether turbinate reduction increases CPAP use or efficacy; and
3. Determine whether turbinate reduction positively influences CPAP treatment outcomes.

We will employ a single-site, randomized, double-blind, sham-placebo-controlled trial to test the hypotheses that turbinate reduction:

1. increases nasal airway cross-sectional area;
2. increases mean nightly objective CPAP use; and
3. improves sleep apnea quality of life 3 months after CPAP titration.

We will use the radiofrequency turbinate reduction surgical technique, which allows ethical randomization and effective blinding. Three, six, and 12 months after turbinate reduction and CPAP titration we will measure the change in the minimal nasal cross-sectional area, level of CPAP use, and improvement in sleep apnea quality of life. Secondary outcomes will capture this treatment's broader impact on the nose, CPAP, and sleep apnea. If turbinate reduction can be shown to improve sleep apnea outcomes through increased use or efficacy of CPAP therapy, this trial will demonstrate the value and effectiveness of a novel, multidisciplinary, combined medical-surgical approach to the management of obstructive sleep apnea syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years
* Newly diagnosed obstructive sleep apnea (apnea-hypopnea index >= 5 events/hour)
* CPAP therapy recommended
* Persistent bilateral inferior turbinate hypertrophy
* American Society of Anesthesiologists Class I-III
* Ability to give informed consent
* Ability and willingness to complete the study protocol
* Fluency in verbal and written English

Exclusion Criteria:

* Previous surgical turbinate treatment
* Other nasal disorders (i.e. recurrent epistaxis, desiccated or crusted mucosa, severe bilateral obstructing septal deformity, or obstructing polyposis)
* Active respiratory tract infections
* Coagulopathy
* Severe psychiatric comorbidity (taking anti-psychotic medication)
* American Society of Anesthesiologists Class IV or V
* Pregnancy
* No telephone
* Plans of moving during the study period
* Known contraindication to lidocaine with epinephrine, oxymetazoline, or acetaminophen

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2007-07; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Nasal minimum cross-sectional area (measured objectively with acoustic rhinometry) | Primary outcome at 3 months, secondary outcomes at 6 and 12 months
CPAP use (measured objectively as pressure-on use) | Primary outcome at 3 months, secondary outcomes at 6 and 12 months
Sleep Apnea Quality of Life Index (change measured with Then Test technique) | Primary outcome at 3 months, secondary outcomes at 6 and 12 months

SECONDARY OUTCOMES:
Secondary Nasal Outcome Measures: peak inspiratory flow, resistance (rhinomanometry), endoscopy, smell identification test, nasal obstruction symptom evaluation (NOSE) scale, and other nasal treatment history | 3, 6, and 12 months
Secondary CPAP Outcome Measures: acceptance, subjective tolerance, pressure, leak, residual breathing events (measured by CPAP device) | 3, 6, and 12 months
Secondary Clinical Outcome Objective Measures: vigilance (psychomotor vigilance task monitor), blood pressure, and plasma C-reactive protein (cardiovascular risk biomarker) | 3, 6, and 12 months
Secondary Clinical Outcome Subjective Measures: Quality of Life Change, Symptoms of Nocturnal Obstruction & Related Events (SNORE-25) Scale, Pittsburgh Sleep Quality Index, Epworth Sleepiness Scale, and Short Form-36 version 2 | 3, 6, and 12 months
Adverse events | Any time research participant reports and scheduled evaluations at 3, 6, and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Edward M. Weaver, MD, MPH, Principal Investigator — University of Washington
Locations (3):
- United States (3):
  - UW Sleep Disorders Center at Harborview Medical Center, Seattle, Washington
  - Virginia Mason Medical Center, Seattle, Washington
  - University of Washington General Clinical Research Center, Seattle, Washington

REFERENCES:
- [Background] Powell NB, Zonato AI, Weaver EM, Li K, Troell R, Riley RW, Guilleminault C. Radiofrequency treatment of turbinate hypertrophy in subjects using continuous positive airway pressure: a randomized, double-blind, placebo-controlled clinical pilot trial. Laryngoscope. 2001 Oct;111(10):1783-90. doi: 10.1097/00005537-200110000-00023. PMID 11801946
- [Background] Li HY, Engleman H, Hsu CY, Izci B, Vennelle M, Cross M, Douglas NJ. Acoustic reflection for nasal airway measurement in patients with obstructive sleep apnea-hypopnea syndrome. Sleep. 2005 Dec;28(12):1554-9. doi: 10.1093/sleep/28.12.1554. PMID 16408415
- [Background] Sugiura T, Noda A, Nakata S, Yasuda Y, Soga T, Miyata S, Nakai S, Koike Y. Influence of nasal resistance on initial acceptance of continuous positive airway pressure in treatment for obstructive sleep apnea syndrome. Respiration. 2007;74(1):56-60. doi: 10.1159/000089836. Epub 2005 Nov 18. PMID 16299414
- [Background] Lam DJ, James KT, Weaver EM. Comparison of anatomic, physiological, and subjective measures of the nasal airway. Am J Rhinol. 2006 Sep-Oct;20(5):463-70. doi: 10.2500/ajr.2006.20.2940. PMID 17063739
- [Background] Stewart MG, Witsell DL, Smith TL, Weaver EM, Yueh B, Hannley MT. Development and validation of the Nasal Obstruction Symptom Evaluation (NOSE) scale. Otolaryngol Head Neck Surg. 2004 Feb;130(2):157-63. doi: 10.1016/j.otohns.2003.09.016. PMID 14990910
- [Background] Friedman M, Tanyeri H, Lim JW, Landsberg R, Vaidyanathan K, Caldarelli D. Effect of improved nasal breathing on obstructive sleep apnea. Otolaryngol Head Neck Surg. 2000 Jan;122(1):71-4. doi: 10.1016/S0194-5998(00)70147-1. PMID 10629486
- [Background] Hilberg O, Pedersen OF. Acoustic rhinometry: recommendations for technical specifications and standard operating procedures. Rhinol Suppl. 2000 Dec;16:3-17. PMID 11225287
- [Background] Flemons WW, Reimer MA. Development of a disease-specific health-related quality of life questionnaire for sleep apnea. Am J Respir Crit Care Med. 1998 Aug;158(2):494-503. doi: 10.1164/ajrccm.158.2.9712036. PMID 9700127
- [Background] Flemons WW, Reimer MA. Measurement properties of the calgary sleep apnea quality of life index. Am J Respir Crit Care Med. 2002 Jan 15;165(2):159-64. doi: 10.1164/ajrccm.165.2.2010008. PMID 11790647
- [Background] Yokoe T, Minoguchi K, Matsuo H, Oda N, Minoguchi H, Yoshino G, Hirano T, Adachi M. Elevated levels of C-reactive protein and interleukin-6 in patients with obstructive sleep apnea syndrome are decreased by nasal continuous positive airway pressure. Circulation. 2003 Mar 4;107(8):1129-34. doi: 10.1161/01.cir.0000052627.99976.18. PMID 12615790
- [Derived] Jara SM, Hopp ML, Weaver EM. Association of Continuous Positive Airway Pressure Treatment With Sexual Quality of Life in Patients With Sleep Apnea: Follow-up Study of a Randomized Clinical Trial. JAMA Otolaryngol Head Neck Surg. 2018 Jul 1;144(7):587-593. doi: 10.1001/jamaoto.2018.0485. PMID 29800001